CLINICAL TRIAL: NCT06683885
Title: A Prospective Clinical Study of the Combination Therapy of Obutinib or Decitabine with Rituximab, Cyclophosphamide, and Prednisone for the Primary Treatment of Elderly Patients with Newly Diagnosed Diffuse Large B-cell Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mingzhi Zhang (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLBCL20141010
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Newly Diagnosed Diffuse Large B-cell Lymphoma
Keywords: DLBCL; clinical trial; chemotherapy; PFS; ORR; Obutinib; Decitabine
MeSH Terms: interventions — Decitabine; Rituximab; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Elderly patients with newly diagnosed DLBCL (Experimental): Obutinib or Decitabine with Rituximab, Compound Cyclophosphamide Tablets and Prednisone
  Interventions: Drug: Obutinib or Decitabine, Rituximab, Compound Cyclophosphamide Tablets and Prednisone

INTERVENTIONS:
Drug: Obutinib or Decitabine, Rituximab, Compound Cyclophosphamide Tablets and Prednisone — For non GCB type: Rituximab, 375mg/m2, QD, D1,8,15(the first cycle), d1(Starting from the second cycle), ivgtt; Compound Cyclophosphamide Tablets, 50mg:50mg BID, P.O.; Obutinib, 150mg, QD, P.O.; Prednisone, 60mg, QD D1-7, P.O. Every 21 days is a cycle, and the efficacy is evaluated every 2 cycles. Obutinib maintain treatment for 6 months. Obutinib, 150mg, QD, P.O. After 6 cycles of initial treatment, the efficacy was evaluated.
  For GCB type: Rituximab, 375mg/m2, QD, D1,8,15(the first cycle), d1(Starting from the second cycle), ivgtt; Compound Cyclophosphamide Tablets, 50mg:50mg BID, P.O.; Decitabine, 10mg, QD，D1-5, ivgtt; Prednisone, 60mg, QD D1-7, P.O. Every 21 days is a cycle, and the efficacy is evaluated every 2 cycles. Decitabine maintenance treatment for 4 cycles, 21 days per cycle. Decitabine, 10mg, QD，D1-5, ivgtt. Evaluate the efficacy after 6 cycles of treatment.

SUMMARY:
A Prospective Clinical Study of the Combination Therapy of Obutinib or Decitabine with Rituximab, Cyclophosphamide, and Prednisone for the Primary Treatment of Elderly Patients with newly Diagnosed Diffuse Large B-cell Lymphoma

DETAILED DESCRIPTION:
This study adopts an open, single arm, prospective clinical collaborative research approach. And the aim is to observe the efficacy and safety of the combination therapy of Obutinib or Desitabine with Rituximab and Cyclophosphamide in elderly patients with newly diagnosed diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 65 years or older who are intolerant to chemotherapy, regardless of gender;
2. ECOG 0-1； IPI score ≤ 3 points;
3. Expected survival period of more than 3 months;
4. DLBCL diagnosed by tissue biopsy pathology;
5. No contraindications for chemotherapy (blood and physiological examination results within 7 days), absolute neutrophil count ≥ 1.0 × 10 ^ 9/L, PLT ≥ 75 × 10 ^ 9/L, hemoglobin ≥ 80g/L (excluding patients with lymphoma bone marrow infiltration);
6. According to the RECIST criteria, there must be at least one measurable lesion. For intranodal lesions, it is defined as: long diameter ≥ 1.5cm and short diameter ≥ 1.0cm; For extranodal lesions, the length and diameter should be ≥ 1.0cm;
7. Liver function: TBIL ≤ 1.5 × ULN; ALT or AST ≤ 2.5 × ULN; Non bone invasive patients with alkaline phosphatase ≤ 3 × ULN;
8. Renal function: serum creatinine ≤ 1.5 × ULN;
9. No other serious illnesses that conflict with this plan;
10. Excluding other major illnesses, the heart function is normal;
11. There are no other related treatments including traditional Chinese medicine (anti-tumor effects), immunotherapy, or biologic therapy (except for treatment of bone metastasis and other symptoms);
12. The subjects voluntarily participate in the clinical trial, sign an informed consent form, and cooperate with follow-up;
13. During this treatment period, if other anti-tumor drugs are not used simultaneously, bisphosphonates can be used for bone metastasis treatment and other symptomatic treatments;

Exclusion Criteria:

1. Clear patients with neurological or psychiatric disorders, including dementia or seizures, a history of abuse of psychotropic drugs that cannot be quit, or other substantial lesions that may increase central neurotoxicity;
2. Individuals who are currently participating in other clinical trials or have participated in other clinical studies within the first 4 weeks of enrollment (excluding those who have not received treatment);
3. Systemic autoimmune diseases or immunodeficiency;
4. Refusing to collect blood samples;
5. Allergic to any medication in the plan;
6. Pregnant and lactating women;
7. Major diseases that can cause experimental interference and uncontrolled active infections;
8. Primary or secondary central tumors;
9. Chemotherapy contraindications;
10. Within 28 days of using Rituximab/Obutinib/Compound Cyclophosphamide Tablets/Azacitidine;
11. Researchers believe that it is not suitable for inclusion;
12. Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infections (excluding nail bed skin fungal infections) or any major systemic infection requiring intravenous antibiotic treatment or hospitalization within the 4 weeks prior to enrollment (excluding tumor fever);
13. Apply other anti-tumor treatments (such as radiotherapy, chemotherapy, hormone therapy, biotherapy, immunotherapy);
14. Other serious diseases that may restrict the subjects from participating in the test, such as uncontrollable diabetes; Severe heart failure (NYHA grade II or above); Acute coronary syndrome has occurred within the past 6 months; Coronary revascularization such as stent implantation, coronary artery bypass surgery, and other heart and large vessel related surgeries within the past 6 months; Severe arrhythmias include frequent premature ventricular contractions, ventricular tachycardia, rapid atrial fibrillation/flutter, and severe bradycardia. Uncontrolled hypertension: systolic blood pressure>150mmHg, diastolic blood pressure>100mmHg. Gastric ulcer (determined by researchers to have a risk of perforation); Active autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia, etc.); Severe respiratory diseases (such as obstructive pulmonary disease and history of bronchospasm), etc;
15. Individuals with bloodthirsty cell syndrome;
16. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) is positive and the detection of hepatitis B virus (HBV) DNA titer in peripheral blood is not within the normal reference value range; Individuals with positive hepatitis C virus (HCV) antibodies and positive hepatitis C virus (HCV) RNA in peripheral blood; Individuals who are HIV antibody positive; Individuals who test positive for Cytomegalovirus (CMV) DNA; Individuals who test positive for syphilis.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | two years
  Overall Response Rate
Progression Free Survival (PFS) | two years
  Progression Free Survival

SECONDARY OUTCOMES:
Overall Survival (OS) | two years
  Overall Survival
Disease free survival（DFS） | two years
  Disease free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Department of The First Affilliated Hospital of Zhengzhou University, Zhengzhou, Henan, China